CLINICAL TRIAL: NCT05763433
Title: Evaluation of Intraoperative Dexamethasone Efficacy to Prevent Rebound Pain Phenomenon According to Individual Patient Characteristics
Brief Title: Variation in the Effect of Dexamethasone Associated With Axillary Plexus on the Occurrence of Rebound Pain
Acronym: VEDR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/28SEP/358
Record Dates: First submitted 2023-01-17; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Adjuvants, Anesthesia; Brachial Plexus Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ambulatory upper limb bone surgery carried out under axillary PNB: Patients will receive a slow intravenous injection of 0.1mg/kg max 10 mg intravenous dexamethasone in a 2cc syringe (5 mg/cc dexamethasone) after PNB is performed, prior to tourniquet placement and the start of surgery.
  Interventions: Other: upper extremity bone surgery

INTERVENTIONS:
Other: upper extremity bone surgery — any ambulatory upper limb bone surgery carried out under axillary PNB

SUMMARY:
The study will evaluate pain and recovery after a single injection axillary plexus block combined with an intravenous dose of 0.1 mg/kg dexamethasone in ambulatory patients undergoing upper extremity bone surgery. The investigators will try to identify the risk factors involved in a decrease in the efficacy of dexamethaxone for the prevention of RP.

The hypotheses are that :

* The interindividual variability may modulate the preventive effect on "rebound pain" after axillary block, of pre-incisional administration of an anti-inflammatory dose of dexamethasone (0.1 mg/kg max 10 mg).
* Patients with increased preoperative anxiety or underlying catastrophizing will experience more postoperative pain as the axillary PNB dissipates.
* Elevated preoperative salivary lipocortin 1 and cortisol levels result in a lesser preventive effect of dexamethasone on the development of rebound pain.

DETAILED DESCRIPTION:
The use of a peripheral nerve block (PNB) through local anesthetics administered may exacerbate the acute inflammatory process induced by the surgical trauma, which may cause rebound pain once the block is lifted, also called "Rebound pain" (RP).

The administration of a dose of Dexamethasone (DEXA) IV as an adjuvant, to optimize the effectiveness of PNB by increasing the duration of PNB , is already a validated practice in anesthesia. In addition the well known analgesic effects of DEXA on postoperative pain (dose> 0.1 mg/kg) seem to contribute to the decrease in RP occurring in the first 24 hours after surgery . These protective properties of DEXA with respect to this phenomenon of hyperalgesia could be explained, among other things, by its modulatory actions on the inflammatory reaction and inhibitory actions on cyclooxygenase as well as its effect on the production of specific mediators such as cytokines.

However, even if DEXA can reduce the onset of RP in some patients, its efficacy seems to be variable and inconsistent between individuals, as suggested by the results of a retrospective observational study .

It can thus be assumed that some individuals are less sensitive to the preventive administration of DEXA and this for different reasons that it would be interesting to better understand .

Objectives:The primary objective will be to identify factors predisposing to variations in the efficacy of DEXA on the occurrence of RP by characterizing the basal stress state of the patient, the level of anxiety and pre-existing catastrophism, as well as the basal thresholds of Lipocortin 1 and cortisol and the basal inflammatory degree (CR high sensitivity) The secondary objective will be to evaluate the interindividual variability of the preventive efficacy of pre-incisional systemic administration of an anti-inflammatory dose of DEXA (0.1 mg/kg, 10 mg maximum) on the occurrence of RP during axillary block removal.

Method: Patients scheduled for elective upper extremity surgery will receive an axillary nerve block. An intravenous injection of DEXA 0.1mg/kg preoperatively will be offered to all patients included in the study. The PNB will be performed under real-time ultrasound guidance by a competent anesthesiologist using a local anesthetic solution of MEPIVACAINE 1%, for volumes administered varying between 15 and 30 ml (maximum 400 mg, 5-6 mg/Kg). The intensity, the neuropathic or catastrophic character of the pain as well as the preoperative anxiety will be collected through specific questionnaires (APAIS /Catastrophisation /CSI /NLR...). In addition, salivary samples of free cortisol and Lipocortin 1 and blood samples (CRP hs and NLR) will be collected before the PNB is performed. All patients will receive, if necessary, an adapted analgesia in the postoperative period and in the recovery room. Patients will be discharged with a standardized analgesic treatment. Patients will be followed up according to the study protocol established in the PACU (recovery room) at D1 to D4 D30 and at 3 months postoperatively (by telephone calls).

ELIGIBILITY:
Inclusion Criteria:

* Any ambulatory upper limb bone surgery carried out under axillary PNB
* Patient aged between 18 and 75 yrs old

Exclusion Criteria:

* Refusal to participate
* Contraindication to the use of Dexamethasone
* Patient with corticoids intake for various reasons
* Contraindication to regular use of postoperative analgesics like non-steroidal anti-inflammatory drugs and paracetamol
* Pregnant woman
* Diabetic patient
* Vascular patient
* Cognitive disorders
* Inability to answer perioperative questionnaires (language problem)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any ambulatory upper limb bone surgery carried out under axillary PNB
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Impact of sexe on the efficacy of DEXA on the occurrence of RP | Through study completion, an average of 1 year
  - Sexe (male ,female),
Impact of BMI on the efficacy of DEXA on the occurrence of RP | Through study completion, an average of 1 year
  - Body mass index BMI (combination of weight measurement in Kilograms and height in meters to obtain BMI in kg/m^2),
Impact of preoperative anxiety levels on the efficacy of DEXA on the occurrence of RP | Through study completion, an average of 1 year
  - Preoperative anxiety levels (APAIS scale). The score can range from 6 ("no anxiety") to 30 ("very anxious").
Impact of preoperative levels of pre-existing catastrophizin on the efficacy of DEXA on the occurrence of RP | Through study completion, an average of 1 year
  - Preoperative levels of pre-existing catastrophizing .(13 items scored from 0 to 4)
Impact of preoperative levels of central sensitization on the efficacy of DEXA on the occurrence of RP | Through study completion, an average of 1 year
  - Preoperative levels of central sensitization index (CSI) (9 questions)
Impact of baseline levels of Lipocortin 1 and cortisol on the efficacy of DEXA on the occurrence of RP | Through study completion, an average of 1 year
  - Baseline levels of Lipocortin 1 and cortisol (salivary assays in nmol/L) and measurements of blood mediators of inflammation, C-Réactive Proteine (CRP) value (in milligrams/liter) and NLR value (neutrophil to lymphocyte ratio) .

SECONDARY OUTCOMES:
Inter-individual variability of preventive efficacy of DEXA | Through study completion, an average of 1 year
  The investigators wish to demonstrate inter-individual variability in the incidence of pain rebound despite systemic pre-incisional preventive administration of an anti-inflammatory dose of DEXA (0.1 mg/kg, 10 mg maximum) for all patients included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nassim TOUIL, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barry GS, Bailey JG, Sardinha J, Brousseau P, Uppal V. Factors associated with rebound pain after peripheral nerve block for ambulatory surgery. Br J Anaesth. 2021 Apr;126(4):862-871. doi: 10.1016/j.bja.2020.10.035. Epub 2020 Dec 31. PMID 33390261
- [Background] Touil N, Pavlopoulou A, Barbier O, Libouton X, Lavand'homme P. Evaluation of intraoperative ketamine on the prevention of severe rebound pain upon cessation of peripheral nerve block: a prospective randomised, double-blind, placebo-controlled study. Br J Anaesth. 2022 Apr;128(4):734-741. doi: 10.1016/j.bja.2021.11.043. Epub 2022 Feb 23. PMID 35219449
- [Background] Stubbs DJ, Levy N. Role of dexamethasone in reducing postoperative pain. Comment on Br J Anaesth 2021; 126: 862-71. Br J Anaesth. 2021 Apr;126(4):e139-e140. doi: 10.1016/j.bja.2021.01.010. Epub 2021 Feb 13. No abstract available. PMID 33589229
- [Background] Desai N, El-Boghdadly K, Albrecht E. Peripheral nerve blockade and novel analgesic modalities for ambulatory anesthesia. Curr Opin Anaesthesiol. 2020 Dec;33(6):760-767. doi: 10.1097/ACO.0000000000000928. PMID 33027077
- [Background] Holmberg A, Hassellund SS, Draegni T, Nordby A, Ottesen FS, Gulestol A, Raeder J. Analgesic effect of intravenous dexamethasone after volar plate surgery for distal radius fracture with brachial plexus block anaesthesia: a prospective, double-blind randomised clinical trial. Anaesthesia. 2020 Nov;75(11):1448-1460. doi: 10.1111/anae.15111. Epub 2020 May 30. PMID 32472958
- [Background] Lavand'homme P. Rebound pain after regional anesthesia in the ambulatory patient. Curr Opin Anaesthesiol. 2018 Dec;31(6):679-684. doi: 10.1097/ACO.0000000000000651. PMID 30124544
- [Derived] Touil N, Pavlopoulou A, Barbier O, Libouton X, Gruson D, Gala JL, Lavand'homme P. Factors associated with a reduction in the preventive effect of intravenous dexamethasone on rebound pain after axillary brachial plexus block. Br J Anaesth. 2025 Oct;135(4):1059-1066. doi: 10.1016/j.bja.2025.05.055. Epub 2025 Jul 22. PMID 40701886